CLINICAL TRIAL: NCT01800162
Title: Optimal Treatment for Women With a Persisting Pregnancy of Unknown Location -- a Randomized Clinical Trial of Women at Risk for an Ectopic Pregnancy
Brief Title: RCT for Women With a Persisting Pregnancy of Unknown Location
Acronym: PPUL
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: A new protocol was written to replace this protocol.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 815013
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2017-12-29 (Actual); Status verified 2017-12

CONDITIONS: Persistent Pregnancy of Unknown Location; Ectopic Pregnancy
MeSH Terms: conditions — Pregnancy, Ectopic | interventions — Methotrexate; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Uterine evacuation, then MTX for some (Active Comparator): Subjects will undergo a uterine evacuation. If hCG levels do not sufficiently decrease after the uterine evacuation, the subject will be treated with methotrexate. If hCG levels do sufficiently decrease after the uterine evacuation, no further treatment is required.
  Interventions: Drug: Methotrexate; Procedure: Uterine Evacuation
- Empiric treatment with MTX for all (Active Comparator): Subjects will be treated with methotrexate, receiving one dose on day 0 and a subsequent dose on day 4. Additional doses will be administered as needed based on hCG levels.
  Interventions: Drug: Methotrexate
- Expectant Management (Active Comparator): Subjects will have their PPUL expectantly managed using serum hCG monitoring.
  Interventions: Other: Expectant Management

INTERVENTIONS:
Drug: Methotrexate — Two Dose Protocol: The patient will receive the first dose of MTX 50mg/m2 on treatment day 0. She will receive a second dose of MTX 50mg/m2 on treatment day 4 and a serum hCG level will be drawn. Subsequent doses of MTX will be administered based on hCG levels.
  Arms: Empiric treatment with MTX for all; Uterine evacuation, then MTX for some
Procedure: Uterine Evacuation — Uterine evacuation or dilation and curettage. At the clinician's discretion, this can be performed using local anesthesia, sedation or general anesthesia and can use a manual or electrical evacuation.
  Arms: Uterine evacuation, then MTX for some
Other: Expectant Management — Pregnancy will be expectantly managed using serum hcg monitoring.
  Arms: Expectant Management

SUMMARY:
This is a randomized controlled trial to compare three currently available management strategies for women with a persisting pregnancy of unknown location (PPUL), which makes them at-risk for ectopic pregnancy. We will recruit hemodynamically stable women with a confirmed PPUL to be randomized to one of three strategies: 1) Uterine evacuation followed by methotrexate (MTX) for some (those that have evidence of a non visualized ectopic pregnancy) 2) Empiric treatment with MTX for all, and 3) Expectant management. Randomization will be 2:2:1 into these three arms. After randomization, they will be followed and treated clinically as is indicated by the progression of their condition. Primary outcome measures: uneventful decline of hCG to 5 IU/mL. Secondary outcome measures: re-interventions, treatment complications, health-related quality of life, financial costs, future fertility, and patient's preferences.

ELIGIBILITY:
Inclusion Criteria:

1. Female with a persisting pregnancy of unknown location:

   1. A pregnancy of unknown location is defined as a women with a positive pregnancy test but no definitive signs of pregnancy in the uterus or adnexa on ultrasound imaging (Ultrasound must be performed within 7 days prior to randomization)
   2. Persistence of hCG is defined as 3 serial hCG values over 4-14 days or 2 serial hCG values over 7-14 days, showing less than 30% rise, or less than 30% fall between the first and last value. (This abnormal pattern of serial hCG confirms that the gestation is nonviable.)
2. Patient is hemodynamically stable, hemoglobin greater than 10 mg/dL,
3. Greater than or 18 years of age

Exclusion Criteria:

1. Hemodynamically unstable in need of acute treatment
2. Most recent hCG greater than 5000 IU/mL
3. Patient obtaining care in relation to a recently completed pregnancy (delivery, spontaneous or elective abortion),
4. Diagnosis of gestational trophoblastic disease,
5. Subject unwilling or unable to comply with study procedures,
6. Presence of clinical contraindications for treatment with methotrexate (ACOG guidelines, Appendix B),
7. Prior medical or surgical management of this gestation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt T Barnhart, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Hospital System University Medical Center, Greenville, South Carolina

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the study has closed at both study sites, The University of Pennsylvania and Greenville.
Pre-assignment Details: Subjects must be 18 years or older. Subject must have a positive pregnancy test but no signs of pregnancy visualized in the uterus or adnexa on ultrasound? Subject must have at least three serial hCG values over the past 4-14 days or two serial hCG values over the past 7-14 days.
  Subject must be hemodynamically stable with a hemoglobin >10mg/dL.
Period: Overall Study
Arm/Group | Uterine Evacuation, Then MTX for Some | Empiric Treatment With MTX for All | Expectant Management
Started (Study ended early only 1 subject randomized to uterine evacuation.) | 1 (1 subject was randomized to uterine evacuation on 6/26/2013.) | 0 | 1 (1 subject randomized to expectant management on 11/1/2013.)
Completed | 1 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uterine Evacuation, Then MTX for Some | Empiric Treatment With MTX for All | Expectant Management | Total
Number analyzed (Participants) | 1 | 0 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1 | 2
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 2
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 0 |  | 1 | 1
  United States | 1 |  | 0 | 1
Gestational Age [Number; unit: weeks] | 14 |  | 7 | 21

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Clinical Resolution for the 3 Different Management Arms for a Persisting PUL.
Description: Data was not analyzed as the study was closed early. Data is not anticipated to be analyzed for this study. Patients were not followed for outcome.
Time Frame: Outcome will be assessed within 6 weeks of randomization
Population: Data was not analyzed as the study was closed early. Data is not anticipated to be analyzed for this study. Patients were not followed for outcome.
Groups:
- Uterine Evacuation; Expectant Management: Data was not analyzed as the study was closed early. Data is not anticipated to be analyzed for this study. Patients were not followed for outcome.
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Ruptured Ectopic Pregnancies in Each Group
Description: as for outcome 1
Time Frame: Outcome will be assess within 6 weeks of randomization
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quantification of Re-interventions Needed to Manage a Woman With a PPUL
Description: Outcomes include:
  * number of interventions beyond that of intended initial strategy in each group
    * additional number of MTX injections
    * additional surgical procedures
  * uterine evacuation (or dilation and curettage)
  * laparoscopy
  * laparotomy
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Treatment Complications and Adverse Events
Description: as for outcome 1
Time Frame: 42 days after the last dose of study medication
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Procedures (Lab Tests, Ultrasounds)
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Visits
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Time to Resolution
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Patients' Preferences
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Acceptability
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation | Expectant Management
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Future Fertility
Description: as for outcome 1
Time Frame: 6 weeks
Arm/Group | Uterine Evacuation, Then MTX for Some | Expectant Management
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- Uterine Evacuation; Expectant Management: No AE to Report
Arm/Group | Uterine Evacuation | Expectant Management
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No